CLINICAL TRIAL: NCT01809184
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0148-0000-0287 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1956-4014; 2012-003048-66 (EudraCT Number); U1111-1132-1018 (Other: WHO)
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Dose level 1 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo
- Dose level 2 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo
- Dose level 3 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo
- Dose level 4 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo
- Dose level 5 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo
- Dose level 6 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo
- Dose level 7 (Experimental): Each subject will be randomly assigned to receive either insulin 287, placebo or insulin glargine within the dose group.
  Interventions: Drug: insulin 287; Drug: insulin glargine; Drug: placebo

INTERVENTIONS:
Drug: insulin 287 — Orally administered insulin 287. The subjects will be dosed in the fasting state and receive one single dose followed by a 24-hour euglycaemic glucose clamp.
Drug: insulin glargine — Insulin glargine administered subcutaneously (s.c., under the skin) at fixed dose levels.
Drug: placebo — Oral placebo adminstered corresponding to insulin 287 treatment

SUMMARY:
This trial is conducted in Europe. The aim of this first human dose trial is to investigate the safety, tolerability, pharmacodynamic (the effect of the investigated drug on the body) and pharmacokinetic (exposure of the trial drug in the body) properties of NNC0148-0000-0287 (insulin 287) in a GIPET® I tablet formulation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0-28.0 kg/m^2
* Subject who is considered to be healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as randomised
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) within 2 weeks prior to dosing, as judged by the investigator
* Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2013-09-06 (Actual); Study Completion 2013-09-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | As recorded from trial product administration and until completion of Sub-visit 2G (Day 13)

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve | From 0 to 648 hours after a single dose
Area under the glucose infusion rate (GIR)-time curve | From 0 to 24 hours after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com